CLINICAL TRIAL: NCT03850197
Title: Comparison of Tubomanometry and EarPopper Devices for Eustachian Tube Function Testing in Children and Adults
Brief Title: Tubomanometry and EarPopper Devices for Eustachian Tube Function Testing
Status: Completed | Type: Observational
Sponsor: Cuneyt M. Alper (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Cuneyt M. Alper, Professor of Otolaryngology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO18050569; P50DC007667 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Eustachian Tube Dysfunction
Keywords: Tubomanometry; EarPopper; Eustachian tube function test
MeSH Terms: interventions — Acoustic Impedance Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TMM followed by EarPopper + Tympanometry: Participants will be asked to complete the tubomanometry (TMM) then EarPopper plus tympanometry tests for each ear, followed by video otoscopy. Nasal endoscopy will also be performed on adult subjects to visualize Eustachian tube (ET) pharyngeal opening and the functional anatomy of surrounding structures during maneuvers. These maneuvers include swallowing, "Fish" maneuver, and blowing out into the EMST-150, and are used to elevate the soft palate to trigger an ET opening.
  Interventions: Device: EarPopper; Device: Tympanometry; Device: Tubomanometry
- EarPopper + Tympanometry followed by TMM: Participants will be asked to complete the EarPopper plus tympanometry then TMM tests for each ear, followed by video otoscopy. Nasal endoscopy will also be performed on adult subjects to visualize ET pharyngeal opening and the functional anatomy of surrounding structures during maneuvers. These maneuvers include swallowing, "Fish" maneuver, and blowing out into the EMST-150, and are used to elevate the soft palate to trigger an ET opening.
  Interventions: Device: EarPopper; Device: Tympanometry; Device: Tubomanometry

INTERVENTIONS:
Device: EarPopper — The EarPopper is 510(K) regulated (510(K) Number K073401) and is marketed as a safe and effective way to aid muscle-assisted ET opening. It is a Politzer device, and aids ET opening by blowing a constant stream of air into the nasal cavity. It consists of a single nose piece connected to an air pump with no adjustable pressure settings. During the study, the subject will be asked to place the nose piece into one of the nostrils while occluding the contralateral. The subject will then perform the maneuvers (swallow, "Fish", blowing out into the EMST-150).
Device: Tympanometry — The Tympanometer is 510(K) regulated (510(K) Number K083861) and is marketed as a way to measure auditory impedance and acoustics reflex by producing controlled levels of test tones and signals. It will be used before and after each maneuver for both the EarPopper and Tubomanometry tests to assess middle ear pressure change.
Device: Tubomanometry — Tubomanometry is an established test of Eustachian tube function. It is an easily-administered test used in clinical laboratories. It consists of a nosepiece and an ear canal pressure probe coupled to a manometer and air pump. When the nosepiece and ear canal probe is in place, a maneuver, such as swallowing, will cause the tubomanometer to generate a bolus of air at 30, 40, or 50 mbar through the nosepiece. In the event that the Eustachian tube opens, the tympanic membrane will be displaced, which in turn will be sensed by the ear probe. This event will be recorded as a Eustachian tube opening. For this test, the investigators will ask the subject to perform the maneuvers (swallow, "Fish", blowing out into the EMST-150).

SUMMARY:
The Eustachian tube (ET) is a biological tube that links the middle ear to the back of the nose and throat. It has several functions, of which the most important is to maintain optimal middle-ear health. Eustachian tube dysfunction (ETD) can result in pain or a popping sensation in the ears when flying in an airplane or going up a tall building in an elevator. Many people with ETD also suffer from ear problems such as repeated middle-ear infections or fluid in the ears. However, there are very few easily-administered tests to measure and assess Eustachian tube function (ETF). Tubomanometry is one of these tests, however it is expensive and used to measure ETF only in research settings. In this study, the investigators propose that using a combination of two readily available devices, the EarPopper and a tympanometer, will work in a manner similar to a Tubomanometer to test ET function.

DETAILED DESCRIPTION:
There is no current universally-accepted set of functional tests or scoring systems for the diagnosis of ETD or measure of the pressure-regulating function of the ET; current practice shows that the diagnosis of ETD relies largely on clinical observation. Though there are several tests that have been developed to characterize ETF, many of them require specialized equipment and trained personnel to administer the test, which are only available in specialized testing centers. As such, this study aims to compare the use of the EarPopper plus tympanometry to Tubomanometry as a ETF test.

Tubomanometry is a simple in-office test based on the Politzer maneuver, in which air is blown into one of the nostrils while occluding the contralateral nostril and swallowing. The tubomanometer consists of an air pump attached to a manometer to adjust the target pressure, a two-pronged nose piece to deliver a controlled airflow to the nostrils and an external ear canal sensor to detect displacement of the tympanic membrane (TM). Since the middle ear is a closed system, displacement of the TM during a swallow is considered a successful ET opening. Tubomanometry is easily tolerated by both adults and children is currently used most widely to evaluate ETF changes after ET balloon dilation. The EarPopper is, like the tubomanometer, a modified politzer device and is used as a treatment device for ET obstruction. It introduces a continuous airflow into the nostril and has no external ear canal probe. The user perceives the ET opening as a subjective sensation of ear fulness. In this pilot study, the investigators will test the feasibility of a new ETF test protocol that will use the EarPopper to trigger the opening of the ET followed by a tympanogram to confirm if there was a change in middle ear pressure. The investigators expect that the combination of these two devices will be comparable to the Tubomanometry test, which will also be performed in the same test session.

Previous studies show that ET opening efficiency is determined by the coordinated function of paratubal muscles, especially of the levator (mLVP) and tensor veli palatini (mTVP) muscles. Nasal endoscopy video recordings have shown a large variability in soft palate closure, as it depends largely on individual effort. For this reason, besides swallowing, the investigators will also employ two additional methods to standardize the elevation of the soft palate and facilitate the opening of the ET: the Fish maneuver (puffing the cheeks and blowing out against a closed mouth) and the EMST-150 device (blowing into the device with a preset low and high resistances). As part of the development of this new testing protocol, these three maneuvers will be used during the EarPopper plus tympanometry and Tubomanometry tests. They will be performed during the EarPopper test, with concurrent video-otoscopy recordings to detect movement of the tympanic membrane that could be interpreted as an ET opening, and during trans-nasal video-endoscopy to record the movement and positioning of the soft palate.

The investigators expect that, in comparing the maneuvers performed during EarPopper plus tympanometry and Tubomanometry tests, they will assess the feasibility of the protocol, define maneuvers to standardize paratubal muscular contraction and determine if the EarPopper plus tympanometry measurements are comparable to Tubomanometry.

ELIGIBILITY:
INCLUSION CRITERIA

ETD participants:

* Bilaterally intact tympanic membranes
* aged 5 to 60; generally good health
* ability to understand and give informed consent
* history of myringotomy tubes, recurrent middle ear infections, recurrent middle ear fluids, or prior ETD diagnosis
* ability to perform maneuvers that will be done during the testing protocol.

Control participants

* Bilaterally intact tympanic membranes
* aged 5 to 60
* generally good health
* ability to understand and give informed consent
* no personal history of recurrent otitis media or other middle--ear disease
* ability to perform maneuvers that will be done during the testing protocol
* no difficulty equalizing middle--ear pressures in daily life.

EXCLUSION CRITERIA

ETD participants:

* Cold/allergic rhinitis (temporary) on presentation
* current dental problem or dental work within 7 days (temporary)
* history of ossicular reconstruction
* history of tympanoplasty
* syndromes predisposing to otitis media
* extant middle--ear disease
* inability to complete testing protocols
* tympanic membrane perforation
* abnormal tympanogram (type B tympanogram)
* BMI >40
* history of congenital heart disease
* prior radiation to head and neck
* uncontrolled respiratory disease
* any medical condition or use of medication for which the study physician feels study procedures would not be in the subject's best interest.
* In adults, a positive urine pregnancy test (in females), blood pressure above 140/90, glaucoma, and sensitivity to drugs used to prepare the nose for endoscopic examination will also exclude potential participants.

Control participants:

* (in addition to above) significant middle--ear disease history
* evidence of middle ear pathology.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 10 healthy adults (aged 18-60), 5 healthy children (aged 5-17), 10 otherwise healthy adults with ETD (aged 18-60), and 5 otherwise healthy children with ETD (aged 5-17) with bilaterally intact TM's will be enrolled after obtaining informed consent. Complete histories will be taken with a focus on any ear-related problems.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Middle ear pressure change after a swallow | Immediately before/after swallow
  The subject's middle ear pressure will be measured before and after they are asked to swallow, while doing the tubomanometry or the Earpopper test. An increase in approximately 10daPa will be considered a Eustachian tube opening.

SECONDARY OUTCOMES:
Middle ear pressure change after "Fish" maneuver | Immediately before/after "Fish" maneuver
  The subject's middle ear pressure will be measured before and after they are asked to carry out the "Fish" maneuver, while doing the tubomanometry or the Earpopper test. An increase in approximately 10daPa will be considered a Eustachian tube opening. The "Fish" maneuver is an effort-dependent method of elevating the soft palate, and will provide further qualitative data on Eustachian tube function.
Middle ear pressure change after blowing into EMST-150 | Immediately before/after blowing into EMST-150
  The subject's middle ear pressure will be measured before and after they are asked to blow out against different levels of resistance into the EMST-150, while doing the tubomanometry or the Earpopper test. An increase in approximately 10daPa will be considered a Eustachian tube opening. Blowing into the EMST-150 is a standardized method of elevating the soft palate, and will provide further qualitative data on Eustachian tube function.

OTHER OUTCOMES:
Movement of tympanic membrane during a swallow | Immediately before/after swallow
  Video otoscopy will be done while subject undergoes the EarPopper plus tympanometry test; movement of the tympanic membrane during a swallow will indicate Eustachian tube opening.
Soft palate elevation to 50% or more of the visual field in 0-degree nasal endoscopy during "Fish" maneuver. | Immediately before/after "Fish" maneuver
  Rigid nasal endoscopy with 0-degree scope will be done on adult subjects while they perform the "Fish" maneuver. Soft palate elevation to 50% or more of the visual field is postulated to be a function of efficient eustachian tube function.

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- ENT Pressure Chamber Laboratory, Oakland Medical Building, 3420 Fifth Avenue, Room 118, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schilder AG, Bhutta MF, Butler CC, Holy C, Levine LH, Kvaerner KJ, Norman G, Pennings RJ, Poe D, Silvola JT, Sudhoff H, Lund VJ. Eustachian tube dysfunction: consensus statement on definition, types, clinical presentation and diagnosis. Clin Otolaryngol. 2015 Oct;40(5):407-11. doi: 10.1111/coa.12475. No abstract available. PMID 26347263
- [Background] Ars B, Dirckx JJJ. Tubomanometry. In: Ars B, ed. Fibrocartilaginous Eustachian Tube-Middle ear cleft. The Hague, The Netherlands: Kugler Publications; 2003:151-158.
- [Background] Esteve D. Tubomanometry and Pathology. In: Ars B, ed. Fibrocartilaginous Eustachian Tube - Middle Ear Cleft. The Hauge, The Netherlands: Kugler Publications; 2003:159-175.
- [Background] Smith ME, Zou CC, Baker C, Blythe AJC, Hutchinson PJA, Tysome JR. The repeatability of tests of eustachian tube function in healthy ears. Laryngoscope. 2017 Nov;127(11):2619-2626. doi: 10.1002/lary.26534. Epub 2017 Feb 22. PMID 28224679
- [Background] Gurtler N, Husner A, Flurin H. Balloon dilation of the Eustachian tube: early outcome analysis. Otol Neurotol. 2015 Mar;36(3):437-43. doi: 10.1097/MAO.0000000000000631. PMID 25356762
- [Background] Schroder S, Lehmann M, Ebmeyer J, Upile T, Sudhoff H. Balloon Eustachian tuboplasty: a retrospective cohort study. Clin Otolaryngol. 2015 Dec;40(6):629-38. doi: 10.1111/coa.12429. PMID 25867023
- [Background] Sheer FJ, Swarts JD, Ghadiali SN. Finite element analysis of eustachian tube function in cleft palate infants based on histological reconstructions. Cleft Palate Craniofac J. 2010 Nov;47(6):600-10. doi: 10.1597/09-131. Epub 2010 Mar 10. PMID 20500073
- [Background] Alper CM, Teixeira MS, Swarts JD, Doyle WJ. Quantitative description of eustachian tube movements during swallowing as visualized by transnasal videoendoscopy. JAMA Otolaryngol Head Neck Surg. 2015 Feb;141(2):160-8. doi: 10.1001/jamaoto.2014.3002. PMID 25474183